CLINICAL TRIAL: NCT04621994
Title: Cesarean Wound Closure: Dermabond Versus Steri Strips
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Laura Grese Willingham, Assistant Professor, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-07302-FB
Record Dates: First submitted 2020-10-30; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steri Strips Arm (Active Comparator)
  Interventions: Other: Steri Strips
- Dermabond Arm (Experimental)
  Interventions: Other: Dermabond

INTERVENTIONS:
Other: Dermabond — Dermabond will be applied after subcuticular skin closure in lieu of Steri Strips
  Arms: Dermabond Arm
Other: Steri Strips — Steri Strips will be applied after subcuticular skin closure as routinely done at our institution
  Arms: Steri Strips Arm

SUMMARY:
The purpose of this study is to determine overall patient satisfaction with their cesarean section scar with application of Steri-strips vs. Dermabond following subcuticular skin closure of pfannenstiel incision

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-45 who are undergoing planned or unscheduled cesarean section at Regional One Health
* Gestational age > 24 weeks
* Planned Pfannenstiel incision
* Willing to consent to the study

Exclusion Criteria:

* Emergency or urgent cesarean section
* Vertical skin incision
* Intrapartum intraamniotic infection
* Diabetes
* Unwilling to consent to the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale Surveys (POSAS) | at 1 weeks postpartum
  Validated scale comparing a scar to normal skin. Score ranges from 6 to 60 with the higher numbers less like normal skin.
Patient and Observer Scar Assessment Scale Surveys | at 6 weeks postpartum
  Validated scale comparing a scar to normal skin. Score ranges from 6 to 60 with the higher numbers less like normal skin.

SECONDARY OUTCOMES:
Number of patients with wound infection | through 6 weeks postpartum
Number of patients with wound separation or dehiscence | through 6 weeks postpartum

IPD SHARING:
Plan to Share IPD: No